CLINICAL TRIAL: NCT05598827
Title: To Observe a Single-center, Randomized, Controlled Clinical Study on the Effect of Douyin on the Emotions of Patients With Bone and Soft Tissue Malignant Tumors During Perichemotherapy
Brief Title: Application of Douyin in Patients With Bone and Soft Tissue Malignant Tumors During Perichemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Jiaqiang, associate chief physician, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZZUSC-15
Record Dates: First submitted 2022-10-23; First posted 2022-10-28 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-11

CONDITIONS: Malignant Tumor; Chemotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Watch the Tik Tok (Experimental): Unlimited Tik Tok viewing was encouraged from 24 hours before chemotherapy until the seventh day after chemotherapy.
  Interventions: Other: Tik Tok
- Tik Tok is not allowed (No Intervention): Viewing of Tik Tok was prohibited from 24 hours before chemotherapy until the seventh day after chemotherapy.

INTERVENTIONS:
Other: Tik Tok — The enrolled patients were encouraged to watch Tik Tok without limit starting 24 days before chemotherapy and continuing until the seventh day after chemotherapy.
  Arms: Watch the Tik Tok

SUMMARY:
A total of 90 patients with bone and soft tissue malignancies who planned to receive chemotherapy were enrolled in this study in Henan Cancer Hospital. They were divided into experimental group and control group for anxiety and depression value 24 hours before chemotherapy, anxiety and depression value on the day of chemotherapy, anxiety value and depression value 24 hours after chemotherapy. To evaluate the effects of watching Tik Tok on perichemotherapy anxiety and depression in patients with bone and soft tissue malignant tumors who were to receive chemotherapy, and to evaluate the effects of watching Tik Tok on the incidence of chemotherapy-related complications in patients with bone and soft tissue malignant tumors who were to receive chemotherapy.

DETAILED DESCRIPTION:
A total of 90 patients with bone and soft tissue malignancies who were scheduled to receive chemotherapy were enrolled in this study in Henan Cancer Hospital. They were divided into experimental group and control group: experimental group: Patients enrolled in this study were encouraged to watch Tik Tok without limit from 24 hours before chemotherapy to the seventh day after chemotherapy. Control group: Viewing Tik Tok was forbidden from 24 hours before chemotherapy to the seventh day after chemotherapy. Anxiety and depression 24 hours before chemotherapy, anxiety and depression 24 hours after chemotherapy, and anxiety and depression 24 hours after chemotherapy. To evaluate the effects of watching Tik Tok on perichemotherapy anxiety and depression in patients with bone and soft tissue malignant tumors who were to receive chemotherapy, and to evaluate the effects of watching Douyin on the incidence of chemotherapy-related complications in patients with bone and soft tissue malignant tumors who were to receive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Men and women aged 10-70. The Eastern Collaborative Oncology Group (ECOG) physical status score was 0-1. Subjects with amputation can be relaxed up to 2 points.

Pathological diagnosis of bone and soft tissue malignancy. Patients who have received at least one previous chemotherapy and are planning to receive new chemotherapy.

All acute toxicities from previous antitumor therapy or surgery resolved to grade 0-1 (according to NCI-CTCAE, version 4.03) or to enrollment/exclusion criteria by day 1 of the first cycle (C1D1), with the exception of toxicities such as hair loss that the investigator considered to pose no safety risk to the subject).

Adequate organ and bone marrow function, as defined below:

Blood routine (no blood transfusion, no G-CSF, no medication correction within 7 days before screening) :

Neutrophil count (ANC)≥1,500/mm3(1.5×109/L); Platelet count (PLT)≥100,000/mm3(100×109/L); Hemoglobin (Hb)≥9g/dL(90g/L);

Blood biochemical:

Serum creatinine (Cr)≤1.5× upper limit of normal (ULN) or creatinine clearance (Cockroft-Gault formula)≥60ml/min; Total bilirubin (TBIL)≤1.5×ULN; Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels ≤2.5×ULN, and subjects with liver metastases should ≤5×ULN;

Blood coagulation function:

International normalized ratio (INR)≤1.5, prothrombin time (PT) and activated partial thromboplastin time (APTT)≤1.5×ULN; With my consent and signed informed consent, I am willing and able to comply with the planned visit, study treatment, laboratory tests and other test procedures.

Exclusion Criteria:

Received the following treatment within 7 days before C1D1:

Radiotherapy, chemotherapy, immune or molecularly targeted therapy for tumors. Some other investigational drugs. Surgery for other sites and/or radiotherapy were planned during the study period (24 hours before chemotherapy and 7 days after chemotherapy).

Imaging diagnosis showed the presence of central nervous system tumor lesions. The presence of active heart disease in the 6 months before C1D1, including myocardial infarction, severe/unstable angina pectoris, etc. Poorly controlled arrhythmias with left ventricular ejection fraction <50% on echocardiography (including QTcF interval >450ms in men and >470ms in women).

In the judgment of the investigator, there are concomitant diseases (such as severe diabetes, neurological or psychiatric diseases) or any other conditions that seriously endanger the safety of the subjects, may confuse the results of the study, or affect the completion of the study.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-28 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety and depression | 24 hours before chemotherapy
  Hospital Anxiety Depression Scale
Anxiety and depression | 1 day of chemotherapy
  Hospital Anxiety Depression Scale
Anxiety and depression | 24 hours after chemotherapy
  Hospital Anxiety Depression Scale

IPD SHARING:
Plan to Share IPD: No